CLINICAL TRIAL: NCT03126929
Title: Further Psychometric Data for the Reliability and the Diagnostic Validity of the Coma Recovery Scale-Revised
Brief Title: Further Psychometric Data for the Reliability and the Diagnostic Validity of CRS-R
Status: Completed | Type: Observational
Sponsor: Hangzhou Normal University (Other)
Responsible Party: Principal Investigator, Ying Zhang, nurse-in-charge, Hangzhou Normal University
Other Study IDs: 2012/026/B
Record Dates: First submitted 2017-04-17; First posted 2017-04-25 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Minimally Conscious State; Vegetative State
Keywords: disorders of consciousness; Vegetative state; Minimally conscious state; Emergence from MCS; Coma Recovery Scale-Revised
MeSH Terms: conditions — Persistent Vegetative State; Consciousness Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Vegetative state: patients lack awareness of self and environment even in the presence for eye-opening and sleep-wake cycles using CRS-R and GCS
  Interventions: Diagnostic Test: Coma Recovery Scale-Revised and Glasgow Coma Scale
- Minimally conscious state: Patients display inconsistent, but reproducible and discernible signs of awareness using CRS-R and GCS
  Interventions: Diagnostic Test: Coma Recovery Scale-Revised and Glasgow Coma Scale
- Emergence from MCS: Patients regain accurate communication and/or functional use of objects using CRS-R and GCS
  Interventions: Diagnostic Test: Coma Recovery Scale-Revised and Glasgow Coma Scale

INTERVENTIONS:
Diagnostic Test: Coma Recovery Scale-Revised and Glasgow Coma Scale — Patients have been assessed with both the Coma Recovery Scale-Revised(CRS-R) and the Glasgow Coma Scale(GCS)

SUMMARY:
This study aims to provide, in a large sample, further psychometric data as regards the internal consistency, the test-retest reliability and the diagnostic validity of the Coma Recovery Scale-Revised (CRS-R).

DETAILED DESCRIPTION:
Recently, a report of the American Congress of Rehabilitation Medicine aiming to provide a systematic review of behavioral assessment scales for DOC has indicated that, when compared to other scales, the CRS-R meets the highest psychometric standards for the evaluation of severely brain-injured patients and may be used to assess DOC with minor reservations. However, that report mentions few evidences or studies with small sample sizes for some aspects of its reliability and validity such as its internal consistency and its test-retest reliability.The report also states that the diagnostic validity of the CRS-R remains unproven. In this study, the investigators will therefore aim to provide further psychometric data as regards those variables in a large sample of patients with DOC

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years old
* any etiology
* pre-screening performed by the referent physician comforting the presence of a disorder of consciousness in accordance with international diagnostic criteria for VS, MCS or emergence from MCS (EMCS)

Exclusion Criteria:

* neuromuscular blocking agents or sedative drugs administered within the prior 24 hours
* no documented history of a prior coma
* critical illness or unstable medical condition

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators chosen patients with VS, MCS, EMCS
Sampling Method: Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised for assess the level of consciousness | 24 hours(1 day)
  Rater Measured the score of Coma Recovery Scale-Revised(CRS-R) within 24h. The CRS-R consists of 23 items grouped in six subscales addressing auditory, visual, motor, oromotor, communication and arousal functions. The lowest item on each subscale represents reflexive activity while the highest items represent cognitively-mediated behaviors.

IPD SHARING:
Plan to Share IPD: Yes